CLINICAL TRIAL: NCT04137341
Title: A Randomized, Open-label, Four-period, Single-dose Cross-over Study in Healthy Male Subjects to Assess the Relative Bioavailability of Two Candidate Tablet Formulations Versus the Current Tablet Formulation of GLPG1972 and to Assess the Food Effect of the Tablet Formulation Selected for Phase 3 in Period 4
Brief Title: A Study in Healthy Volunteers to Compare Different Tablet Formulations of the Test Medicine, GLPG1972, Against the Current Tablet Formulation, and to Assess the Effect Food Has on One of the Test Medicines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG1972-CL-109; 2019-002144-25 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tablet A (Experimental): A single oral 300-mg dose of GLPG1972 in fasted state
  Interventions: Drug: GLPG1972 - A
- Tablet B (Experimental): A single oral 300-mg dose of GLPG1972 in fasted state
  Interventions: Drug: GLPG1972 - B
- Tablet C (Experimental): A single oral 300-mg dose of GLPG1972 in fasted state
  Interventions: Drug: GLPG1972 - C
- Food effect (Experimental): selected tablet B or C under fed conditions
  Interventions: Drug: GLPG1972 - B; Drug: GLPG1972 - C

INTERVENTIONS:
Drug: GLPG1972 - A — Film-coated tablet, formulation A
  Arms: Tablet A
Drug: GLPG1972 - B — Film-coated tablet, formulation B
  Arms: Food effect; Tablet B
Drug: GLPG1972 - C — Film-coated tablet, formulation C
  Arms: Food effect; Tablet C

SUMMARY:
The sponsor wants to investigate two new tablet formulations (recipes) of the test medicine, and how they are taken up by the body in comparison to the current tablet formulation (study periods 1 to 3). If one of the 2 new tablets has a more favourable profile than the current tablet in periods 1 to 3, the sponsor will then investigate the effect that food has on this new tablet in study period 4. However, if the new tablets do not have a more favourable profile than the current tablet, the food effect does not need to be investigated and study period 4 will not be needed.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18-55 years of age (extremes included), on the date of signing the informed consent form
* A body mass index (BMI) between 18.0-30.0 kg/m2, inclusive
* Judged to be in good health by the investigator based upon the results of medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests. Clinical laboratory safety test results must be within the reference ranges or considered not clinically significant in the opinion of the investigator
* Subject must be able and willing to comply with restrictions on prior medication as described in the protocol
* Negative screen for drugs (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants) and alcohol

Exclusion Criteria:

* Known hypersensitivity to IMP ingredients or history of a significant allergic reaction to the investigational medicinal product (IMP) ingredients as determined by the investigator, and/or known sensitivity to IMP or the excipients (e.g. lactose). Hay fever is allowed unless active.
* Positive serology for hepatitis B virus surface antigen or hepatitis C virus or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first IMP administration.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus infection)
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first IMP administration.
* Presence or sequelae of gastrointestinal, liver, kidney (creatinine clearance ≤80 mL/min, using the Cockcroft-Gault formula: if calculated result is ≤80 mL/min, a 24-hour urine collection can be done) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero until the time corresponding with the last observed quantifiable concentration calculated by the linear up (AUC0-t) ratio between tablet formulations | From Day 1 pre-dose up to Day 4
  To assess the bioavailability of two candidate tablet formulations (Tablet B and Tablet C) relative to that of the current tablet formulation (Tablet A) of GLPG1972
Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) ratio between tablet formulations | From Day 1 pre-dose up to Day 4
  To assess the bioavailability of two candidate tablet formulations (Tablet B and Tablet C) relative to that of the current tablet formulation (Tablet A) of GLPG1972
Maximum observed plasma concentration (Cmax) ratio between tablet formulations | From Day 1 pre-dose up to Day 4
  To assess the food effect of the selected Phase 3 tablet formulation (in case Tablet B or Tablet C) of GLPG1972
Area under the plasma concentration-time curve from time zero until the time corresponding with the last observed quantifiable concentration calculated by the linear up (AUC0-t) ratio between fed and fasted | From Day 1 pre-dose up to Day 4
  To assess the food effect of the selected Phase 3 tablet formulation (in case Tablet B or Tablet C) of GLPG1972
Area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) ratio between fed and fasted | From Day 1 pre-dose up to Day 4
  To assess the food effect of the selected Phase 3 tablet formulation (in case Tablet B or Tablet C) of GLPG1972
Maximum observed plasma concentration (Cmax) ratio between fed and fasted | From Day 1 pre-dose up to Day 4
  To assess the bioavailability of two candidate tablet formulations (Tablet B and Tablet C) relative to that of the current tablet formulation (Tablet A) of GLPG1972

SECONDARY OUTCOMES:
The number of incidents of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs) and TEAEs leading to discontinuations | From Day 1 through study completion, an average of 2 months
  To evaluate the safety and tolerability of oral doses of GLPG1972 tablet formulations

CONTACTS AND LOCATIONS:
Overall Officials: Angela de Haas-Amatsaleh, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Limited, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No